CLINICAL TRIAL: NCT04802928
Title: Healing of Ischemic Leg Ulcers: A Pilot Trial
Brief Title: Healing of Ischemic Leg Ulcers in Patients Treated With iSONIAzid
Acronym: SONIA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Patients fulfilling the criteria could not be found.
Sponsor: Pharma 2100 (Industry)
Responsible Party: Principal Investigator, Magnus Agren, Professor, Pharma 2100
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007-003387-22
Record Dates: First submitted 2008-03-31; First posted 2021-03-17 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Arterial Leg Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Placebo Comparator): Placebo tablets.
  Interventions: Drug: Placebo
- B (Experimental)
  Interventions: Drug: Isoniazid 300 milligram

INTERVENTIONS:
Drug: Isoniazid 300 milligram — Tablets 150 milligram b.i.d.
  Arms: B
Drug: Placebo — Placebo
  Arms: A

SUMMARY:
The main objective of this trial is to study the healing effect of an oral drug (isoniazid) in patients with ischemic (arterial) leg ulcers defined by a systolic toe pressure <40 mm Hg.

DETAILED DESCRIPTION:
Treatment of arterial ulcers is problematic. Previous pharmaceutical interventions with for example prostaglandins have produced only limited beneficial effects but have been associated with frequent adverse effects. Positive effects of isoniazid have been observed in a preclinical model of ischemic wound healing (Weinreich et al. Surgery 2010).

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic leg ulcers unsuitable for vascular surgical intervention
* Systolic toe pressure < 40 mm Hg
* Ulcer duration > 3 months
* Ulcer area: 1-20 cm2
* Written informed consent

Exclusion Criteria:

* B-Hb < 6 mmol/l
* Aspartate transaminase > 50 U/l
* Diabetes mellitus > 10%HbA1c
* Usage of more than 10 mg prednisolone daily within the last 30 days
* Usage of cytotoxic agents with the last 3 months
* Usage of rifampicin, phenytoin, carbamazepin, theophylline, benzodiazepines (diazepam, triazolam), stavudine and/or valproat
* Alcohol abuse
* Hereditary galactose intolerance
* Hypersensitive to isoniazid or for one or more of the filling substances (magnesium stearate, povidone, talcum, lactose and starch)
* Cellulitis or deep infection (osteomyelitis and/or tendonitis) related to the ulcer
* Gangrene
* Participation in clinical trials within the last 7 days
* Pregnancy or breastfeeding
* Women of child bearing potential who decline to use contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2008-09 (Estimated); Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
The percentage change of ulcer area 8 weeks after initiation of therapy. | 8 weeks
  The wound area is measured at week 0 (A0) and at 8 weeks (A8). From these measurements, the percentage (%) change of the wound area in relation to the start time (week 0) is determined from the following formula: (A0-A8)/A0*100.

SECONDARY OUTCOMES:
Pain is evaluated by visual analogue scale (VAS). | 8 weeks
  The visual analogue scale ranges from 0 mm (minimum) to 100 mm (maximum), where the lower value the better is the outcome.
Occurrence of suspected unexpected serious adverse reactions (SUSAR) and serious adverse events (SAE) | 8 weeks
  the number of SUSAR and SAE occurring over the 8-week treatment period is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Tonny Karlsmark, MD, PhD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark